CLINICAL TRIAL: NCT06668155
Title: Isolated Autograft Anterior Cruciate Ligament Reconstruction Versus Allograft Anterior Cruciate Ligament Reconstruction With Lateral Extra-articular Tenodesis: A Randomized Controlled Trial
Brief Title: ACLR: Isolated Autograft vs Allograft With Lateral Extra-articular Tenodesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amit Momaya, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300012655; UAB (Other: UAB)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: ACL Deficient Knee
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: * Assignment 0 represents the autograft group. If assigned the autograft group, the surgeon will choose either bone patella tendon bone (BPTB) or all soft tissue quadriceps tendon for the graft. The graft choice will be based upon surgeon preference.
  * Assignment 1 represents allograft with lateral extra-articular tenodesis LET group. The allograft used will be a non-irradiated quadriceps tendon with bone plug allograft with a donor age less than 45 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assignment 0 (Active Comparator)
  Interventions: Procedure: Autograft Group
- Assignment 1 (Active Comparator)
  Interventions: Procedure: Allograft with LET Group

INTERVENTIONS:
Procedure: Autograft Group — If assigned the autograft group, the surgeon will choose either bone patella tendon bone (BPTB) or all soft tissue quadriceps tendon for the graft. The graft choice will be based upon surgeon preference.
  Arms: Assignment 0
Procedure: Allograft with LET Group — The allograft used will be a non-irradiated quadriceps tendon with bone plug allograft with a donor age less than 45 years.
  Arms: Assignment 1

SUMMARY:
This study seeks to evaluate the utility of non-irradiated allograft tissue with lateral extra-articular tenodesis (LET) in the setting of anterior cruciate ligament reconstruction (ACLR).

DETAILED DESCRIPTION:
While ACL injuries are among the most common sports medicine injuries treated arthroscopically, significant debate surrounds the choice of graft used in ACLR. While graft choice has been studied extensively, allografts have been shown to have a slightly increased risk of failure than autografts. However, these differences become less pronounced with non-irradiated allografts that have not undergone chemical processing or with slower rehabilitation timelines. Allografts also show poorer graft maturation on MRI. The use of allografts may avoid the donor site morbidities associated with autograft procedures such as pain, donor site weakness, and increased surgical duration. Previous studies have documented a high prevalence of extensor and flexor weakness following autograft ACLR, with deficits in flexor strength following hamstring autograft lasting up to 12 months and extensor strength deficits at 24 months following quadriceps tendon autograft ACLR. Limiting these morbidities may allow a more predictable return to activity and improve patient satisfaction following ACLR. Despite the benefits, concern remains regarding the use of allografts in higher demand patients. However, some studies of patients undergoing ACLR show similar results between allografts and autografts.

Despite advancements in ACLR techniques, retear rates and return-to-play rates remain unsatisfactory in specific populations. Recent investigations into the persistence of anterolateral rotatory laxity in patients have led to an increased focus on the role of the anterolateral complex for knee stability. Specifically, LET has grown in popularity in the setting of ACLR. Previous studies have demonstrated that the addition of LET may improve clinical outcomes when performed in conjunction with an ACLR, possibly by decreasing post-operative pivot shift, tibial translation, and retear rates.

No study to date has compared non-irradiated allografts augmented with LET to autografts for ACLR in a randomized controlled trial fashion. This proposed study aims to understand the utility of allografts in ACLR when combined with LET.

ELIGIBILITY:
Inclusion Criteria:

* ACL deficient knee that are indicated for autograft ACLR

Exclusion Criteria:

* concomitant ligamentous injury that require surgery
* revision ACLR
* patients indicated for LET
* patients with previous knee surgery
* patients with cancer
* patients who are pregnant or nursing

Ages: 14 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2028-01 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Anterior Tibial Translation | 9 month post procedure
  KT-1000 measurement
Quadricep and Hamstring Strength | 5-8 months post procedure and 9-15 months post procedure
  Isometric Biodex Testing
Magnetic Resonance Imaging | 9-15 months post procedure
  Graft signal interpretation

CONTACTS AND LOCATIONS:
Overall Officials: Amit Momaya, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Undecided